CLINICAL TRIAL: NCT05272618
Title: Clinical Relevance of Coronary Microvascular Dysfunction Assessments in Myocardial Infarction With Non-Obstructive Coronary Arteries
Brief Title: Coronary Microvascular Dysfunction Assessments in Myocardial Infarction With Non-Obstructive Coronary Arteries
Acronym: CMD-MINOCA
Status: Recruiting | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Korean Cardiac Research Foundation (Unknown); Abbott (Industry)
Responsible Party: Principal Investigator, Young Joon Hong, Professor, Chonnam National University Hospital
Other Study IDs: CNUH-2021-413
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction; Coronary Microvascular Dysfunction; Vasospasm, Coronary
Keywords: MINOCA; Coronary physiology; Cardiac PET; CFR; IMR; OCT
MeSH Terms: conditions — Myocardial Infarction; Coronary Vasospasm; MINOCA | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MINOCA with CMD: MINOCA patients with CMD proven by invasive or non-invasive method
  Interventions: Diagnostic Test: Intravascular imaging (OCT), Invasive physiologic assessment (FFR, CFR, IMR), or Non-invasive physiologic assessment (N-13 ammonia PET)
- MINOCA without CMD: MINOCA patients without CMD
  Interventions: Diagnostic Test: Intravascular imaging (OCT), Invasive physiologic assessment (FFR, CFR, IMR), or Non-invasive physiologic assessment (N-13 ammonia PET)

INTERVENTIONS:
Diagnostic Test: Intravascular imaging (OCT), Invasive physiologic assessment (FFR, CFR, IMR), or Non-invasive physiologic assessment (N-13 ammonia PET) — Intravascular imaging (OCT), Invasive physiologic assessment (FFR, CFR, IMR), or Non-invasive physiologic assessment (N-13 ammonia PET)

SUMMARY:
To compare clinical outcomes of myocardial infarction with non-obstructive coronary arteries (MINOCA) according to the coronary microvascular dysfunction (CMD), evaluated by optical coherence tomography (OCT), invasive and non-invasive coronary physiologic assessment.

DETAILED DESCRIPTION:
Background Approximately 5~10% of patients with acute myocardial infarction (AMI) have been reported as myocardial infarction with non-obstructive coronary arteries (MINOCA) in the contemporary clinical setting. Although those with MINOCA have a better prognosis than with obstructive coronary artery disease, several observational studies continuously reported that patients with MINOCA showed comparable outcomes. One plausible explanation of this discrepancy is the heterogeneous and variable definition of MINOCA. Possible causes of MINOCA include plaque erosion and/or rupture, vasospasm, and CMD. Therefore, it is natural that heterogeneous pathophysiology of MINOCA causes diagnostic challenges and proper management.

Recently, there have been efforts for establishing the diagnosis of MINOCA and standardizing the systematic management according to the cause of MINOCA. According to the AHA scientific statement, patients who suspected MINOCA have been recommended to perform multimodality approach, including intravascular imaging (i.e., OCT). Although non-invasive methods, such as N-13 ammonia positron emission tomography (PET), can be used for evaluating the CMD, invasive coronary physiologic assessment using pressure-temperature wire has been recommended. CMD has been known as a major cause of MINOCA, and it may be required specific treatment.

Nevertheless, there has no data on the outcomes of MINOCA with or without CMD. Therefore, the aim of CMD-MINOCA sought to assess the MINOCA patients regarding the latest clinical pathway for diagnosis of CMD and evaluate their clinical outcomes at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age ≥19 years and acute myocardial infarction

  * Rise and/or fall of cardiac troponin with one level >99 percentile plus ischemic signs/symptoms

    * Subject with non-obstructive coronary arteries
  * <50% diameter stenosis or
  * fractional flow reserve (FFR) >0.80 ③ Subject without previous history of coronary artery disease

    * Subject who performed invasive coronary angiography within 24 hours after presentation ⑤ Subject who eligible for invasive and non-invasive coronary physiologic assessment

Exclusion Criteria:

* Subject with obstructive coronary arteries

  * Subject with alternate diagnosis including sepsis, pulmonary embolism, myocarditis, Takotsubo syndrome, spontaneous coronary dissection, and other cardiomyopathies.

    * Subject with cardiogenic shock or cardiac arrest ④ Subject who has non-cardiac co-morbid conditions with life expectancy <1 year ⑤ Subject or lactating women ⑥ Subject unable to provide consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 150 patients with suspected myocardial infarction underwent invasive coronary angiography, but without obstructive coronary arteries will be enrolled. These patients will be evaluated by OCT, coronary functional assessment including coronary spasm test, invasive (FFR, CFR, IMR) and non-invasive coronary physiologic assessment (N-13 ammonia positron emission tomography).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE | 2-Year after enrollment
  a composite of cardiac death, any MI, any revascularization, stroke, readmission due to heart failure

SECONDARY OUTCOMES:
cardiac death | 2-Year after enrollment
  death from cardiac-cause
all-cause death | 2-Year after enrollment
  death from any-cause
Rate of myocardial infarction | 2-Year after enrollment
  any type of myocardial infarction
Rate of repeat revascularization | 2-Year after enrollment
  ischemia-driven or all
Rate of stroke | 2-Year after enrollment
  ischemic or hemorrhagic stroke by brain imaging
re-admission due to heart failure | 2-Year after enrollment
  re-admission due to heart failure
all-cause death, any MI, or any revascularization | 2-Year after enrollment
  a composite of all-cause death, any myocardial infarction, or any revascularization
Changes of left ventricular ejection fraction | 2-Year after enrollment
  left ventricular ejection fraction by echocardiography
Changes of Coronary flow reserve | 6-Month after enrollment
  Coronary flow reserve by PET

CONTACTS AND LOCATIONS:
Overall Officials: Young Joon Hong, MD, PhD, Principal Investigator — Chonnam National University Medical School; Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the main paper, we have a plan to share IPD regarding the request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 31, 2026 ~
Access Criteria: Not specified. To be discussed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT05272618/Prot_SAP_000.pdf